CLINICAL TRIAL: NCT00825110
Title: SS-GCC1- Screening Study of Genetic Changes in Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR3085
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Cancer
Keywords: colorectal; cancer; gene expression; biomarker; genomic mismatch repair
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biospecimen includes formalin-fixed, paraffin embedded tissue, fresh frozen tissue and blood smaples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment: confirmed diagnosis of colorectal carcinoma

SUMMARY:
the principal research objective is to form a database of tissue samples from patients with colorectal (bowel) cancer. The tissue samples that will be used for this research will have already been taken for diagnostic or therapeutic reasons. We will also be asking for consent for a research blood sample. The database will be used to improve our understanding of the molecular genetics and gene expression patterns in colorectal cancer.

DETAILED DESCRIPTION:
All patients at the Royal Marsden with a diagnosis of colorectal cancer will be eligible to enter this study. This will include patients both with early and advanced disease, provided they give informed consent. They will give written consent to participate, to include consent for analysis of existing tumour tissue and consent for collection of demographic and clinicopathological data relating to their case and its future outcome, and consent for a blood sample to be taken for research purposes. Additionally, old samples of material surplus to clinical requirements may be collected without specific consent if there is no possibility that it would affect the patient's interest (eg the patient has died).

ELIGIBILITY:
Inclusion Criteria:

* adults who have a terminal illness
* 18 and over
* confirmed diagnosis of colorectal carcinoma
* ability to give informed consent
* paraffin embedded histological material available for analysis

Exclusion Criteria:

* medical or psychiatric conditions
* impairing ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients at the Royal Marsden with a diagnosis of colorectal cancer will be eligible to enter this study.
  Adults who have a terminal illness
Sampling Method: Probability Sample
Enrollment: 3750 (Estimated)
Dates: Start 2008-11; Primary Completion 2020-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
the primary endpoint is the identification of cases with evidence of loss of the product of one of the four main MMR genes on tumour histology.

SECONDARY OUTCOMES:
Secondary outcome measure is the survival and response to treatment of the identified cases.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Cunningham, David, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom